CLINICAL TRIAL: NCT01019096
Title: Absorption of Heme and Non-Heme Iron in Pregnant and Non-pregnant Women and Mechanisms of Fetal Iron Transfer
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 06-06-045; 2006-07-160 (Other Grant/Funding Number: HATCH, Cornell University)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Iron Deficiency
Keywords: iron; pregnancy; heme iron; non-heme iron; stable isotopes; women/adolescents
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For non-pregnant subjects 15 mL of blood are collected. For pregnant subjects two 15 mL blood samples are collected. The placenta and up to 30 mL of cord blood are also collected at delivery.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The three specific aims of this study are 1) to assess the impact of iron status on relative differences in absorption of heme and non-heme iron among pregnant women and non-pregnant women, 2) to assess the magnitude and the determinants of heme and non-heme iron transfer to the fetus over the last trimester of pregnancy, and 3) to characterize relationships between placental iron binding proteins with the enrichment of stable iron isotopes in the neonate at birth. The investigators hypothesize that there will be up regulation of heme and non-heme iron absorption and up regulation of placental iron transport proteins in response to low maternal iron stores.

DETAILED DESCRIPTION:
To measure the absorption of heme and non-heme iron in women, pregnant and non-pregnant women will consume a standardized meal of pork (intrinsically labeled with 58Fe) and a second meal of non-heme 57Fe (as ferrous sulfate). Two weeks after ingesting these test meals, a blood sample will be collected from each women and the amount of heme (58Fe) and non-heme (57Fe) iron incorporated into red blood cells will be measured with magnetic sector thermal ionization mass spectrometry. Cord blood samples and placental tissue will be obtained at delivery to measure how these two forms of dietary iron were transferred across the placenta to the fetus. Maternal and neonatal iron status and placental proteins involved in iron transport will also be measured. Data from this study will provide information that aims to improve human health by better understanding the iron requirements of a population at high risk of iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant subjects (15-35 yrs): non-smoking,healthy with uncomplicated pregnancies at time of enrollment
* Non-pregnant subjects (18-35 yrs): healthy, non-smoking, not taking vitamin or mineral supplements and not planning on becoming pregnant during course of study.

Exclusion Criteria:

* Pregnant subjects: gestational diabetes, hypertension, preeclampsia, underlying malabsorption diseases or other diagnosed medical problems known to impact iron homeostasis
* Non-pregnant subjects: underlying malabsorption diseases or other diagnosed medical problems known to impact iron homeostasis.

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women and adolescents from Rochester, NY and non-pregnant women from Ithaca, NY.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Heme and Non-Heme Iron Absorption | two-weeks post dosing (3rd trimester for pregnant subjects)
Heme and Non-Heme Transfer to Fetus | Delivery

SECONDARY OUTCOMES:
Iron Status (serum ferritin, TfR, Total Body Iron, Hb, Hepcidin), Folate, B-12, CRP and EPO in women and neonates | two weeks post dosing and at delivery for pregnant subjects
Protein expression of key iron transport proteins. | Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O O'Brien, PhD, Principal Investigator — Cornell University; Eva Pressman, MD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Highland Hospital, Rochester, New York
  - Strong Memorial Hospital, Rochester, New York

REFERENCES:
- [Result] Young MF, Griffin I, Pressman E, McIntyre AW, Cooper E, McNanley T, Harris ZL, Westerman M, O'Brien KO. Maternal hepcidin is associated with placental transfer of iron derived from dietary heme and nonheme sources. J Nutr. 2012 Jan;142(1):33-9. doi: 10.3945/jn.111.145961. Epub 2011 Nov 23. PMID 22113871
- [Result] Young MF, Griffin I, Pressman E, McIntyre AW, Cooper E, McNanley T, Harris ZL, Westerman M, O'Brien KO. Utilization of iron from an animal-based iron source is greater than that of ferrous sulfate in pregnant and nonpregnant women. J Nutr. 2010 Dec;140(12):2162-6. doi: 10.3945/jn.110.127209. Epub 2010 Oct 27. PMID 20980658
- [Result] Young MF, Pressman E, Foehr ML, McNanley T, Cooper E, Guillet R, Orlando M, McIntyre AW, Lafond J, O'Brien KO. Impact of maternal and neonatal iron status on placental transferrin receptor expression in pregnant adolescents. Placenta. 2010 Nov;31(11):1010-4. doi: 10.1016/j.placenta.2010.08.009. Epub 2010 Sep 15. PMID 20828813
- [Derived] Delaney KM, Guillet R, Pressman EK, Caulfield LE, Zavaleta N, Abrams SA, O'Brien KO. Iron absorption during pregnancy is underestimated when iron utilization by the placenta and fetus is ignored. Am J Clin Nutr. 2020 Sep 1;112(3):576-585. doi: 10.1093/ajcn/nqaa155. PMID 32614379